CLINICAL TRIAL: NCT01253941
Title: Effects of Mud Bath Therapy in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, Simonetta Baldi, Dr., Fondazione Salvatore Maugeri
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MBT-COPD2010_FORSTIII; 1050 FoRST (Other Grant/Funding Number: FoRST)
Record Dates: First submitted 2010-12-02; First posted 2010-12-06 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD, Intensive Resistive Breathing, Cytokine IL6,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Mud Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mud Bath therapy (Experimental)
  Interventions: Other: Mud bath Therapy
- no Mud Bath Therapy (No Intervention)

INTERVENTIONS:
Other: Mud bath Therapy — patients will be randomized to Mud bath Therapy ( 12 sessions) or no treatment
  Other Names: Thermal treatment
  Arms: Mud Bath therapy

SUMMARY:
Rehabilitation and physical therapy strategies targeting extra pulmonary manifestations of Chronic Obstructive Pulmonary Disease (COPD)are far from being well defined. Studies, performed in healthy subjects using threshold breathing device [a simple method to increase inspiratory muscle load] have shown that ventilatory muscle overactivation during loaded breathing may prime reactive oxygen species (ROS) production, thus initiating an inflammatory response that results in elevation of pro-inflammatory cytokines, particularly IL_6. Increase of cytokine IL_6 in turn, elicits a cascade of systemic responses, involving hormone like glucoregulatory mechanisms, lipolysis and fat oxidation, as well as control of breathing.

Thermal mud bath therapy has been acknowledged for its antioxidant and anti-inflammatory effects in several chronic diseases. However, it is not considered among treatment options of chronic pulmonary disease. Previous experimental studies indicate that trace elements of thermal treatments, particularly iodide and bromide, may positively intervene in the setup and maintenance of active state in skeletal muscle. These findings suggest that in COPD patients these elements may improve the loading and endurance of respiratory muscles and therefore blunt ventilatory muscle overactivation and the ensuing inflammatory cytokine response.

In this study the investigators want to test two major hypotheses. First, that mud bath therapy reduces systemic inflammatory processes in COPD patients, increases respiratory muscle endurance and normalizes the ventilatory response. Second, that the increase in systemic inflammation after IRB exercise is blunted by mud bath therapy.

DETAILED DESCRIPTION:
The impact of extra pulmonary manifestations of Chronic Obstructive Pulmonary Disease (COPD) on physical performance and quality of life, together with the notion that plasma cytokines in COPD is not due to an overflow of inflammatory mediators from the lung compartment, raise interest in understanding the potential link between lung and systemic inflammation.

Recent studies, performed in normal subjects using threshold breathing device [a simple method to increase respiratory resistance and inspiratory muscle load] have shown that ventilatory muscle activation during loaded breathing may prime reactive oxygen species (ROS) production, thus initiating an inflammatory response within diaphragm that results in systemic elevation of pro-inflammatory cytokines. These findings provide a sound working hypothesis about the origin of systemic inflammation in COPD. Endurance and task failure of inspiratory muscles can be challenged during inspiratory resistive breathing (IRB) exercise performed with either nonlinear or threshold loading devices [4-6], thus allowing to simulate resistive breathing caused by airway narrowing occurring during COPD exacerbations Therapy with mineral water is a widely used modality of physical therapy in countries rich in mineral water. Up to date, however, it is not considered among treatment options of chronic pulmonary disease by recent guidelines. Mud bath therapy has been acknowledged for its antioxidant and anti-inflammatory effects in several chronic diseases. Although full mechanisms of such effects have not yet been fully elucidated, previous in vivo studies on the effects of several anions on the duration of active state in skeletal muscle indicate that trace elements of thermal treatments, particularly iodide and bromide, may positively intervene in the setup and maintenance of this active state. These findings suggest that in COPD patients these elements may improve the loading and endurance of respiratory muscles and therefore blunt ventilatory muscle overactivation and the ensuing inflammatory cytokine response.

In this study the investigators want to test two major hypotheses. First, that mud bath therapy reduces systemic inflammatory processes in COPD patients, increases respiratory muscle endurance and normalizes the ventilatory response. Second, that the increase in systemic inflammation after IRB exercise is blunted by mud bath therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 45 years
* 34% </= FEV1 </= 70%
* stable clinical conditions

Exclusion Criteria:

* idiopathic or acquired bronchiectasis
* cardiovascular, peripheral vascular or cerebrovascular disease
* systemic confounding inflammatory disease (e.g rheumatoid arthritis,Crohn's disease, systemic vasculitis etc.)
* malignancies

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cytokine IL6 at 2weeks +2days (after Mud Bath Therapy) | baseline test before IRB, at Day 17
  Subjects for the study will be 42 mild-to-severe COPD outpatients. They will carry out baseline venous and arterial capillary blood sampling, ventilatory response tests and assessment of pulmonary function, before and after loaded breathing (IRB)test. Patients will then be randomized to standard mud bath therapy (12 sessions) or no-treatment. All tests and measurements will be repeated afterwards.
Change before-after IRB test in cytokine IL_6, at baseline | before-after IRB test, at Day 0
  Subjects for the study will be 42 mild-to-severe COPD outpatients. They will carry out baseline venous blood sampling, before and after loaded breathing (IRB)test. Change before-after IRB test in IL_6 will be assessed at baseline(day 0).
Change before-after IRB test in cytokine IL_6, at 2 weeks +2 days | before-after IRB test, at Day 17
  Subjects for the study will be 42 mild-to-severe COPD outpatients. They will carry out baseline venous blood sampling, before and after loaded breathing (IRB) test. Change before-after IRB test in IL_6 will be assessed again at 2 weeks + 2days(day 17, after Mud Bath Therapy).

SECONDARY OUTCOMES:
Change from baseline in respiratory muscle endurance time, at 2weeks +2days | IRB test duration, at Day 17
  Time duration of sustainable inspiratory pressure, set at 50% of MIP
Change from baseline in Ventilatory Response to CO2, at 2weeks +2days | Baseline test at day 17
  Ventilatory response to CO2 (VRCO2), is conducted according to Read's technique. The subjects will be seated comfortably, attached to the mouthpiece with a noseclip in place and breathing room air until the end-tidal PCO2 (Pet,CO2) stabilized. They then will start rebreathing a mixture of approximately 7% CO2 and 93% O2. Rebreathing was continued for at least 3 minutes.
Change before-after IRB test in VRCO2, at day 0 | before-after IRB test, at Day 0
  Ventilatory response to CO2 (VRCO2), conducted according to Read's technique, will be obtained before and after IRB test, at day 0
Change before-after IRB test in VRCO2, at day 17 | before-after IRB test, at Day 17
  Ventilatory response to CO2 (VRCO2), conducted according to Read's technique, will be obtained before and after IRB test, at day 17

CONTACTS AND LOCATIONS:
Overall Officials: Simonetta Baldi, MD, Principal Investigator — Fondazione Salvatore Maugeri; Gian Domenico Pinna, Ph.D, Principal Investigator — Fondazione Salvatore Maugeri
Locations (2):
- Italy (2):
  - Fondazione Salvatore Maugeri- Istituto Scientifico di Montescano, Montescano, Pavia
  - Salvatore Maugeri Foundation - Scientific Institute of Montescano, Montescano, Pavia

REFERENCES:
- [Result] Vassilakopoulos T, Hussain SN. Ventilatory muscle activation and inflammation: cytokines, reactive oxygen species, and nitric oxide. J Appl Physiol (1985). 2007 Apr;102(4):1687-95. doi: 10.1152/japplphysiol.01273.2006. Epub 2006 Dec 21. PMID 17185492
- [Result] Martyn JB, Moreno RH, Pare PD, Pardy RL. Measurement of inspiratory muscle performance with incremental threshold loading. Am Rev Respir Dis. 1987 Apr;135(4):919-23. doi: 10.1164/arrd.1987.135.4.919. PMID 3565939
- [Result] Nickerson BG, Keens TG. Measuring ventilatory muscle endurance in humans as sustainable inspiratory pressure. J Appl Physiol Respir Environ Exerc Physiol. 1982 Mar;52(3):768-72. doi: 10.1152/jappl.1982.52.3.768. PMID 7068493
- [Derived] Baldi S, Pinna GD, Bruschi C, Caldara F, Maestri R, Dacosto E, Rezzani A, Popovich E, Bellinzona E, Crotti P, Montemartini S, Fracchia C. Medicinal clays improve the endurance of loaded inspiratory muscles in COPD: a randomized clinical trial of nonpharmacological treatment. Int J Chron Obstruct Pulmon Dis. 2015 Oct 23;10:2235-48. doi: 10.2147/COPD.S87999. eCollection 2015. PMID 26604728
- [Derived] Baldi S, Jose PE, Bruschi C, Pinna GD, Maestri R, Rezzani A, Bellinzona E, Fracchia C, Dacosto E, Crotti P, Montemartini S. The mediating role of cytokine IL-6 on the relationship of FEV(1) upon 6-minute walk distance in chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2014 Oct 7;9:1091-9. doi: 10.2147/COPD.S57845. eCollection 2014. PMID 25336940